CLINICAL TRIAL: NCT02257671
Title: The Influence of Oral Contraceptives on Mood, Sexuality and Economic Behavior
Brief Title: Oral Contraceptives and Economic Behaviour
Acronym: P-piller101
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Angelica Lindén Hirschberg, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-020824-23
Record Dates: First submitted 2014-09-28; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Female Contraception
MeSH Terms: interventions — Contraceptives, Oral; Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral contraceptive (Active Comparator): oral dose of ethinylestradiol 0.03 mg + levonorgestrel 0.15 mg per day during 11 weeks
  Interventions: Drug: Oral contraceptive
- Placebo (Placebo Comparator): Oral placebo capsule daily during 11 weeks
  Interventions: Drug: Oral contraceptive

INTERVENTIONS:
Drug: Oral contraceptive — Neovletta
  Other Names: ethinylestradiol + levonorgestrel

SUMMARY:
The investigators aim is to evaluate effects of combined oral contraceptives (OC) on mood, sexuality and economic behaviour in a randomized, double-blind, placebo-controlled study. 400 healthy women will be randomized to OC or placebo for a period of three months. Before and at the end of treatment, mood and sexuality will be assessed by validated instruments. At the end of treatment, each woman will participate in behavioral experiments testing self-confidence, risk taking and altruism. The current project could fill the gap of ignorance about causal effects of OCs on mood, sexuality and behavior. The results might improve current practice as regards information about OCs, choice of hormonal contraceptive, regimen and duration of use. As a consequence, this could lead to reduced discontinuation rate, fewer unintended pregnancies and abortions. The project will contribute to an overall improvement in women's reproductive health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young women, aged 18-35 years, BMI 19-30

Exclusion Criteria:

* Risk factors for thrombosis, smoking, obesity, hypertension, diabetes and estrogen/gestagen therapy the last three months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
economic behaviour | 11 weeks
  A modified dictator game will be used to measure altruistic behavior (Eckel and Grossman 1996). Each subject decides how to allocate money between herself and a charitable organisation. The size of the donation is our measure of altruism. Risk aversion is measured by a test where the subject makes several choices between a certain payoff and a 50/50 gamble to win a certain amount of money (Dohmen et al 2005). Competitiveness is defined as the extent to which women choose to compete in a task which involves solving as many simple mathematical exercises as possible during three minutes (Niederle and Vesterlund 2007).
sexual behaviour | baseline to 11 weeks
  Sexual function will be assessed by the validated instruments Sexual Activity Log (SAL) (Derogatis et al 2004), Profile of Female Sexual Function (PFSF) (McHorney et al 2004, Derogatis et al 2004) and Personal Distress Scale (PDS, past 30 days) (Derogatis et al 2004, Leiblum et al 2006). The women are answering the questionnaires, which are all computerized, at the Women´s Health Research Unit.
mood | baseline to 11 weeks
  Mood and health-related quality of life will be assessed by the Beck Depression Inventory (BDI) test (Lightfoot and Oliver 1985) and the Psychological General Well-Being Index (PGWB) (Dupuy 1984, Wiklund et al 1992).

CONTACTS AND LOCATIONS:
Overall Officials: Angelica L Hirschberg, Professor, Principal Investigator — Department of Obstetrics and Gynecology, Karolinska University Hospital, Stockholm, Sweden
Locations (1):
- Department of Obstetrics and Gynecology, Karolinska University Hospital, Stockholm, Sweden